CLINICAL TRIAL: NCT01977196
Title: Phase 1 of DTP/Hepatitis B 10ug Hib Vaccine
Brief Title: The Safety and Immunogenicity of DTP/Hepatitis B 10ug Hib Vaccine (Bio Farma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Penta 0111
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: DTB/HB/Hib vaccine; Infants; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DTP/HepatitisB/Hib vaccine (Experimental): Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis HbsAg PRP-TT Aluminum phosphate Natrium Chloride Thimerosal
  Interventions: Biological: DPT/HepatitisB/Hib vaccine

INTERVENTIONS:
Biological: DPT/HepatitisB/Hib vaccine — DPT/HepatitisB/Hib vaccine (Bio Farma)
  Other Names: Pentavalent

SUMMARY:
The objective of this study was to know the safety of DTP/Hepatitis B and Hib/PRP-T vaccine and immediate reactions within the first 30 minutes after injection.

DETAILED DESCRIPTION:
This trial was an open-label study, no randomization, and no placebo or control group. Total 30 healthy infants (age 6-11 weeks) followed this trial. The safety was assessed within 24 hours, 48 hours, 72 hours, and 28 days after injection.

ELIGIBILITY:
Inclusion Criteria:

* Infant 6-11 week of age
* Infant born after 37-42 week of pregnancy
* Infant weighting more than 2.5 kg at birth
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form
* Parents commit themselves to comply with the indication of the investigator and with the schedule of the trial

Exclusion Criteria:

* Child concomitantly enroll or schedule to be enroll in another trial
* Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature >=37.5 Celsius on Day 0)
* Known history of allergy to any component of the vaccine component (e.g.formaldehyde)
* History of uncontrolled coagulopathy or blood disorder contraindicating intramuscular injection
* Known history of congenital or acquired immunodeficiency (including HIV infection)
* Child who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived product or long term corticotherapy (>2 minggu)
* Other vaccination within the 7 days prior to inclusion with the exception of BCG and poliomyelitis
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objective
* Infant with a known history of diphteria, tetanus, pertussis, Hib, Hepatitis B infection

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse event of DTP/Hepatitis B/Hib vaccine (Bio Farma) | 30 minutes
  Local and systemic reactions

SECONDARY OUTCOMES:
Incidence rate of adverse event of DTP/Hepatitis B/Hib vaccine (Bio Farma) | 28 hours, 48 hours, 72 hours, 28 days
  Local and systemic reaction
To asses the immunogenicity | 28 days
  Percentage of infants with increasing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, PhD, Principal Investigator — Faculty of Medicine UNPAD
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia